CLINICAL TRIAL: NCT01159834
Title: Proposal for HPV Vaccination of Women in the City of Barretos. A Pioneering Project Designed by the Pio XII Foundation - Barretos Cancer Hospital.
Brief Title: Human Papillomavirus (HPV) Vaccination in Barretos (Pio XII Foundation - Barretos Cancer Hospital)
Status: Completed | Type: Observational
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jose Humberto Tavares Guerreiro Fregnani, PhD, PhD, Barretos Cancer Hospital
Other Study IDs: Vaccine HCB 01
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Human Papillomavirus; Infection
Keywords: HPV infection; Cervical cancer; HPV vaccine
MeSH Terms: conditions — Infections; Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gardasil, HPV infection

SUMMARY:
PROJECT JUSTIFICATION: Cervical cancer is a serious public health problem in Brazil, and is the cause of significant morbidity and mortality among Brazilian women. In spite of government efforts to improve the coverage rates of Pap tests, the disease-related incidence and mortality rates remain high and the diagnosis is still too late.Considering that the chronic human papillomavirus (HPV) related genital infection leads to cervical cancer development, cervical cancer should be the target of primary prevention through vaccination.

PROJECT OBJECTIVES: This project aims to evaluate de following vaccination indicators: 1) Program acceptance rate; 2) Vaccine coverage rate; 3) Three-dose completion rate; 4) Rescue vaccination demand; 5) Adverse event rate;

TARGET POPULATION: Schoolgirls attending the 6th and 7th grades of elementary school (mean age = 11.9 yo).

VACCINATION PROGRAM: The program adopted the quadrivalent vaccine because it is considered superior to the bivalent vaccine in preventing HPV-induced lesions. In addition to preventing the development of pre-cancer lesions and cervical cancer, the quadrivalent vaccine has also proved to be effective in preventing condyloma, and vaginal and vulvar cancer. The girls received the vaccines doses at their schools (school-based program) and also at the Barretos Cancer Hospital.

RESULTS:

Program acceptance rate = 91.8% (95%CI: 87.0%-96.8%);

Vaccine coverage for 1st, 2nd and 3rd doses = 87.5% (95%CI: 82.9%-92.2%), 86.3% (95%CI: 81.8%-91.1%) and 85.0% (95%CI: 80.5%-89.7%).

Three dose completion rate = 97.2% (95%CI: 92.0%-100.0%). Reasons for dropping out of the vaccination program included: moving out of town (17), lost during follow up (16), guardians' decision but without a reasonable justification (3), girl refused to continue in the program (1) and pregnancy (2). Two girls interrupted the vaccination because of adverse events reported by the parents.

Rescue vaccination demand = 279 girls on the first dose (20.3%; 95%CI: 17.9%-22.8%), 357 on the second dose (26.3%; 95%CI=23.6%-29.1%) and 291 on the third dose (21.7%; 95%CI=19.3%-24.4%).

Thirty adverse events were recorded or observed in 4,074 doses, providing an adverse event rate of 0.7% (95%CI: 0.5%-1.1%). There was no severe adverse event.

ELIGIBILITY:
Inclusion Criteria:schoolgirls, attending the 6th and 7th grades of the elementary school.

Exclusion Criteria:Pregnant and breastfeeding adolescents and girls who did not attend classes.

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study included young girls enrolled in public and private schoolgirls, attending the 6th and 7th grades of the elementary school. Pregnant and breastfeeding adolescents and girls who did not attend classes (although enrolled at school) were excluded. Considering the inclusion criteria, 19 schools were candidates to the project (13 public and 6 private). The list provided by each school accounted for 1,615 girls, out of which, 41 were not eligible for the study. Thus, 1,574 girls were considered as potential candidates to the vaccination program.
Sampling Method: Non-Probability Sample
Enrollment: 1574 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José H Fregnani, PhD, Principal Investigator — Barretos Cancer Hospital